CLINICAL TRIAL: NCT03449290
Title: Assistant Professor, Physioterapist, PhD
Brief Title: The Short-term Effects of Trunk Kinesio Taping on Trunk Muscle Endurance and Postural Stability in Healthy Young Adults
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ataturk Training and Research Hospital (Other)
Responsible Party: Principal Investigator, Seyda TOPRAK CELENAY, Assist Prof, PT, PhD, Ataturk Training and Research Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2018-45/48
Record Dates: First submitted 2018-02-17; First posted 2018-02-28 (Actual); Last update posted 2018-02-28 (Actual); Status verified 2018-02

CONDITIONS: Kinesio Taping

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Kinesio taping group (Experimental): Kinesio taping was applied on trunk muscles
  Interventions: Other: Kinesio taping
- Control group (Sham Comparator): Sham Kinesio taping was applied on trunk muscles
  Interventions: Other: Sham Kinesio taping

INTERVENTIONS:
Other: Kinesio taping — Kinesio taping was applied on both sides of rectus abdominus, obliquus internus, obliquus externus and sacrospinalis muscles with muscle technique
  Arms: Kinesio taping group
Other: Sham Kinesio taping — Kinesio taping was applied on both sides of rectus abdominus, obliquus internus, obliquus externus and sacrospinalis muscles without any technique
  Arms: Control group

SUMMARY:
This study aimed to investigate the short-term effects of trunk kinesio taping on trunk muscle endurance and postural stability in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy young volunteers aged between 18-25 years

Exclusion Criteria:

* Having disc hernias, any spinal pain complaint, spinal deformity, history related to spinal surgery, vestibulopathy, musculoskelatal injuries related to ankle, knee and hip joints, orthopedic and/or neurological problems and allergy to the kinesio tape

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2018-02-15 (Actual); Primary Completion 2018-03 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Trunk muscle endurance | Change from Baseline taping at 1 hour after the taping
  Trunk muscle endurance with McGill's trunk muscle endurance tests (seconds) was assessed

SECONDARY OUTCOMES:
Postural stability | Change from Baseline taping at 1 hour after the taping
  Postural stability as static using a force platform when eyes open and eyes closed was assessed

CONTACTS AND LOCATIONS:
Overall Officials: Seyda TOPRAK CELENAY, Study Director — Ankara Yildirim Beyazıt University; Nezehat Ozgul UNLUER, Principal Investigator — Ankara Yildirim Beyazıt University; Taskin OZKAN, Principal Investigator — Ankara Yildirim Beyazıt University
Locations (1):
- Ankara Yildirim Beyazit University, Ankara, Turkey (Türkiye)